CLINICAL TRIAL: NCT06691945
Title: Prophylactic Amnioinfusion for Prevention of Postpartum Hemorrhage: A Randomized Clinical Trial (PURPOSE)
Brief Title: Prophylactic Amnioinfusion for Prevention of Postpartum Hemorrhage
Acronym: PURPOSE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sarah Mehl, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-24-0439
Record Dates: First submitted 2024-11-11; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prophylactic amnioinfusion (Experimental)
  Interventions: Combination Product: Saline delivered using an intrauterine pressure catheter (IUPC)
- Routine Care (No Intervention)

INTERVENTIONS:
Combination Product: Saline delivered using an intrauterine pressure catheter (IUPC) — An intrauterine pressure catheter (IUPC) will be placed in participants after membrane rupture, or at 4 cm if membranes previously ruptured. A 300cc bolus of normal saline will be administered. A continuous rate of 100 cc/hr of normal saline will continue until delivery to prevent Postpartum Hemorrhage. If the IUPC is dislodged, it will be replaced by a trained clinician.
  Arms: Prophylactic amnioinfusion

SUMMARY:
The purpose of this study is to decrease the likelihood of composite postpartum hemorrhage (PPH) morbidity, which consists of i) Estimated or quantified blood loss of 1,500 mL or more, ii) transfusion of any blood products or iii) hysterectomy

ELIGIBILITY:
Inclusion Criteria:

* Singletons with a gestational age of 34.0 weeks or more
* Labor (spontaneous or medical induction)
* Medium- or High-risk for PPH, as described by American College of Obstetricians and Gynecologists (ACOG)

Exclusion Criteria:

* Scheduled cesarean delivery
* Multiple gestations
* Delivery at < 34.0 weeks
* Contraindication to place intrauterine pressure catheter (e.g. HIV)
* Incarcerated subjects
* Major fetal anomalies requiring neonatal surgical intervention
* Stillbirth on admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2026-11-11 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have estimated or quantified blood loss of 1,500 mL or more | from delivery admission to discharge (average of 3 days post delivery)
Number of participants who have transfusion of any blood products | from delivery admission to discharge or up to 12 weeks post delivery
Number of participants who have hysterectomy | from delivery admission to discharge or up to 12 weeks post delivery

SECONDARY OUTCOMES:
Number of mothers who use uterotonics, in addition to oxytocin | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Estimated blood loss(mL) | post delivery (from immediately after delivery to upto 2 hours after delivery)
Quantitative blood loss(mL) | post delivery(from immediately after delivery to upto 2 hours after delivery)
Delta change in hemoglobin of mothers | pre delivery, post partum day 1
Number of mothers who have cesarean deliveries | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of mothers who need Mechanical tamponade | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of mothers who have surgical interventions (O'Leary, B 'Lynch or uterine arterial embolization) | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of mothers who have Chorioamnionitis | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of mothers who have endometritis | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of mothers who have wound complications (if cesarean delivery) | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of mothers who are admitted to intensive care unit | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of deaths | from delivery admission to discharge or up to 12 weeks post delivery if participant is readmitted in the postpartum period
Number of neonates with Apgar < 7 | at 5 minutes after delivery
Number of neonates that have a seizure | delivery admission to discharge or upto 27 days after birth if neonate is readmitted with any of the complications
Number of neonates that have meconium aspiration syndrome | delivery admission to discharge or upto 27 days after birth if neonate is readmitted with any of the complications
Number of neonates that have Ventilation > 6 hrs | delivery admission to discharge or upto 27 days after birth if neonate is readmitted with any of the complications
Number of neonates that have Bronchopulmonary dysplasia | delivery admission to discharge or upto 27 days after birth if neonate is readmitted with any of the complications
Number of neonates that have Necrotizing enterocolitis | delivery admission to discharge or upto 27 days after birth if neonate is readmitted with any of the complications
Number of neonates that have Sepsis | delivery admission to discharge or upto 27 days after birth if neonate is readmitted with any of the complications
Number of stillbirths | at delivery
Number of deaths of neonates | within 27 days of birth

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mehl, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No